CLINICAL TRIAL: NCT00135889
Title: Improving Postoperative Rehabilitation Following Total Knee Arthroplasty With Perineural Local Anesthetic Infusion
Brief Title: Continuous Femoral Nerve Block Following Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Collaborators: Foundation for Anesthesia Education and Research (Other); Arrow International (Industry); Stryker Instruments (Industry); University of Florida (Other); University of California, San Diego (Other)
Responsible Party: Brian M. Ilfeld, MD, MS; Principal Investigator, University of California at San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 560-2003; GCRC 582; GCRC Grant RR00082
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Pain
Keywords: Total Knee Arthroplasty secondary to osteoarthritis
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Femoral perineural infusion

SUMMARY:
The purpose of this study is to determine if putting local anesthetic-or numbing medication-through a tiny tube next to the nerves that go to the knee will improve pain control during physical therapy, and ultimately improve the results of surgery. It will also determine if patients having knee replacement surgery may receive the same or better pain control at home compared with staying in the hospital, and if this improves their experience following surgery.

DETAILED DESCRIPTION:
What procedures would be done as part of your normal clinical care (even if you did not participate in this research)?

You will have some monitors placed (such as a blood-pressure cuff) and be given some medicines through your intravenous (IV) line to make you very sleepy. The anesthesiologist will then place a nerve block so that much of your knee (not all) will be numb. At the same time, the anesthesiologist will place a tiny tube, called a catheter, near your nerves that will be used after the surgery is over. You will still go to sleep for the surgery, but you will be much more comfortable when you wake up because the numbing medicine will be working to take away much of the pain. If you are not part of this study, you would go from the recovery room to a room in the hospital for 3-5 days, and your catheter would be removed the morning following surgery. After your catheter was removed, you would depend on oral and IV opioids-or pain medicine-to control your surgical pain. You would go home with only oral opioids since IV opioids cannot be provided at home.

What procedures will be done only because you are participating in this research study?

From the recovery room you will go to the Clinical Research Center (CRC) which is a special part of the hospital where research is undertaken. During your stay at the CRC you will have the ability to push a button on a small infusion pump to give yourself more medicine through the tube to your nerves if you have pain. If this does not help enough, you will take pain pills to help. And if this does not help enough, you will be given opioids (strong pain medicine like morphine) into your IV. Each morning after surgery, the medicine in your little infusion pump will be replaced by either (1) more medicine, or (2) salt water, or "normal saline". The pharmacist will determine this randomly-like flipping a coin-and neither you nor the doctors/nurses caring for you will know which you have. This is to keep any of us from inadvertently/unconsciously affecting the results of the study. However, if you have pain that is not controlled with pain pills, you will be switched back to the regular medicine to improve your comfort until the following morning. You will undergo physical therapy and following this you will be checked to see if you are ready to go home. When you are ready to go home beginning on the third day after surgery, you may go home with the little infusion pump and the tube that goes to the nerves of your knee. One of the study physicians will call you each night to ensure that you are comfortable for the first 7 nights after your surgery, and you will be given the phone and pager numbers of a physician available for you to contact 24 hours/day, 7 days/week. When the medicine runs out or in the fourth evening following surgery, whichever comes first, your catheter will be removed. The pump is disposable, so it can be thrown away. A physician will call you the two nights after the catheter comes out to ensure that you are comfortable.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral, primary total knee arthropathy (TKA)
* 18-80 years of age
* Be able to understand the possible local anesthetic-related complications, study protocol, and care of the catheter and infusion pump system and are already planning on having a perineural catheter placed for postoperative analgesia

Exclusion Criteria:

* Any contraindication to femoral block/catheter
* Any comorbidity which results in moderate or severe functional limitation (American Society of Anesthesiologists [ASA] physical status >2)
* Baseline oxygen saturation < 96% on room air
* Known hepatic or renal insufficiency (creatinine level > 1.5 mg/dL)
* Allergy to study medications (other than nonsteroidal anti-inflammatory agents [NSAIDs] and acetaminophen)
* Inability to communicate with the authors
* Morbid obesity (body mass index [BMI]>40 kg/m2)
* History of opioid abuse or chronic regular opioid use (use within the 2 weeks prior to surgery and duration of use > 4 weeks)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Distance of ambulation in the afternoon following surgery
Time from surgical stop until three discharge criteria are met

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California San Diego, La Jolla, California
  - University of Florida, Gainesville, Florida

REFERENCES:
- [Background] Ilfeld BM, Gearen PF, Enneking FK, Berry LF, Spadoni EH, George SZ, Vandenborne K. Total knee arthroplasty as an overnight-stay procedure using continuous femoral nerve blocks at home: a prospective feasibility study. Anesth Analg. 2006 Jan;102(1):87-90. doi: 10.1213/01.ane.0000189562.86969.9f. PMID 16368810
- [Result] Ilfeld BM, Le LT, Meyer RS, Mariano ER, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Theriaque DW, Berry LF, Spadoni EH, Gearen PF. Ambulatory continuous femoral nerve blocks decrease time to discharge readiness after tricompartment total knee arthroplasty: a randomized, triple-masked, placebo-controlled study. Anesthesiology. 2008 Apr;108(4):703-13. doi: 10.1097/ALN.0b013e318167af46. PMID 18362603
- [Derived] Ilfeld BM, Meyer RS, Le LT, Mariano ER, Williams BA, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Maldonado RC, Gearen PF. Health-related quality of life after tricompartment knee arthroplasty with and without an extended-duration continuous femoral nerve block: a prospective, 1-year follow-up of a randomized, triple-masked, placebo-controlled study. Anesth Analg. 2009 Apr;108(4):1320-5. doi: 10.1213/ane.0b013e3181964937. PMID 19299806